CLINICAL TRIAL: NCT01339650
Title: A Phase 1 Study of ABT-767 in BRCA1 or BRCA2 Mutation Carriers With Advanced Solid Tumors and in Subjects With High Grade Serous Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Study of ABT-767 in Subjects With Breast Cancer 1 and Breast Cancer 2 (BRCA 1 and BRCA 2) Mutations and Solid Tumors or High Grade Serous Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-976; 2010-020795-37 (EudraCT Number)
Record Dates: First submitted 2011-04-04; First posted 2011-04-21 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Fallopian Tube; Primary Peritoneal Cancer; Solid Tumors (e.g. Breast, Ovarian, Prostate, or Pancreatic) and Ovarian
Keywords: Solid Tumor; BRCA 1 and BRCA 2 Mutations; Breast Cancer 1; Breast Cancer 2; High Grade Serous Ovarian, Fallopian Tube, or Primary Peritoneal Cancers; Solid Tumors
MeSH Terms: conditions — Fanconi Anemia, Complementation Group D1 | interventions — ABT-767

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABT-767 (Experimental): ABT-767 monotherapy
  Interventions: Drug: ABT-767

INTERVENTIONS:
Drug: ABT-767 — ABT-767 once or twice daily for a 28 day cycle

SUMMARY:
This is a Phase 1, dose escalation trial evaluating the tolerability, pharmacokinetics, and pharmacodynamics of ABT-767 in subjects with advanced Breast Cancer 1 or 2 gene (BRCA1 or BRCA2)-mutated solid tumors and high grade serous ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
This is a Phase 1, dose escalation trial evaluating the tolerability, pharmacokinetics, and pharmacodynamics of ABT-767 in subjects with advanced BRCA1 or BRCA2-mutated solid tumors and high grade serous ovarian, fallopian tube, or primary peritoneal cancer. ABT-767 is a potent oral inhibitor of the enzymes poly (ADP-ribose) polymerase 1 and 2 (PARP-1 and PARP-2). Malignancies with deficiencies in homologous repair, such as BRCA-1 and BRCA-2 deficient tumors, are more dependent on PARP for deoxyribonucleic acid (DNA) repair than normal cells and, thus, are thought to be more sensitive to PARP inhibition. The study design is a single-arm dose escalation study to determine dose-limiting toxicities, maximum tolerated dose and the recommended Phase 2 dose (RPTD) of orally administered ABT-767 in subjects with BRCA mutations and malignancies. In order to further evaluate the safety and tolerability of ABT-767 at the RPTD, 20 additional subjects will be enrolled in an expanded safety cohort consisting of BRCA1- or BRCA2-mutated Breast cancer and Ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 years of age.
2. Subjects must have histological or cytological confirmation of locally advanced or metastatic solid tumor, and a documented Breast Cancer Gene 1 or 2 mutation, or high grade serous ovarian, fallopian tube, or primary peritoneal cancer.
3. Subject has an Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 2
4. Subjects must have adequate hematologic, renal, and hepatic function as follows: a. Bone Marrow: Absolute neutrophil count (ANC ≥ 1,500/mm3 (1.5 ≥ 109/L); Platelets ≥ 100,000/mm3 (100 ≥ 109/L); Hemoglobin ≥ 9.0 g/dL (1.4 mmol/L) (hemoglobin unsupported by transfusion b. Subject has adequate renal function as demonstrated by serum creatinine value of ≤ 1.5 x the upper limit of normal (ULN) and either an estimated creatinine clearance value of ≥ 50 mL/min as determined by the Cockcroft-Gault formula or a creatinine clearance value of ≥ 50 mL/min/1.73 m2 based on a 24-hour urine collections c. Subject has adequate liver function as demonstrated by serum bilirubin ≤ 1.5 x ULN and Aspartate Aminotransferase (AST) and Alanine Transaminase (ALT) ≤ 2.5 ULN. For subjects with liver metastasis, AST and ALT < 5 x ULN. Partial Thromboplastin Time (PTT) must be ≤ ULN and INR < 1.5. - Subjects on anticoagulant (such as Coumadin) are allowed on study and will have PTT and International Normalize Ratio (INR) as determined by the Investigator.
5. Women of childbearing potential must agree to use adequate contraception prior to study entry, for the duration of the study participation, and for 90 days following completion of therapy. Women of childbearing potential must have a negative serum pregnancy test within 21 days prior to initiation of treatment and a negative urine pregnancy test on the first day of study drug administration. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria:

1. Expanded cohort only: Subject has previously received a poly (ADP-ribose) polymerase (PARP) inhibitor.
2. Subject has received anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, biologic or any investigational therapy within a period of 28 days or 5 half lives (whichever is shorter) prior to Study Day 1.
3. Subject has known Central Nervous System (CNS) metastases.
4. Subject has unresolved toxicities from prior anti-cancer therapy, defined as any Common Terminology Criteria for Adverse Events (CTCAE v 4.0) grade 2 or higher clinically significant toxicity (excluding alopecia).
5. Subject has had major surgery within 28 days prior to Study Day 1.
6. Clinically significant uncontrolled condition(s) or any medical condition which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities.
7. Psychiatric illness/social situation that would limit compliance with study requirements.
8. Lactating or pregnant female.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-05-06 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile | Various time points from Cycle 1 Day -4 to Day 8
  Blood samples for pharmacokinetics of ABT-767 will be collected at designated time points

SECONDARY OUTCOMES:
Safety (number of subjects with adverse events and/or dose limiting toxicities) | Weekly for the first two months, every other week for the third month, and monthly there after. An expected average is 5 months.
  Adverse events, laboratory results, physical exams and vital signs will be evaluated throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (3):
- Netherlands (3):
  - Univ Med Center Groningen, Groningen
  - Univ Med Ctr, St. Radboud, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam

IPD SHARING:
Plan to Share IPD: No